CLINICAL TRIAL: NCT03613519
Title: Reducing Health Disparities for Black Women in the Treatment of Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-37156; AD-2017C1-6314 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-04

CONDITIONS: Insomnia
Keywords: Patient education; Sleep hygiene; Sleep Healthy Using the Internet (SHUTi); Cognitive-behavioral therapy (CBT); Black Women's Health Study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Hygiene | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomly assigned to one of the 3 intervention groups; SHUTi-BWHS, SHUTi, or patient education (PE).
Who Masked: Participant
Masking Description: Participants do not know the treatment at the time of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient education (sleep hygiene) (Placebo Comparator): A web-based program that presents ways to improve behaviors and environments that can affect sleep.
  Interventions: Behavioral: Patient education
- SHUTi (Sleep Healthy Using the Internet) (Active Comparator): SHUTi is web-based cognitive-behavioral therapy instrument for insomnia (CBT-I)
  Interventions: Behavioral: SHUTi
- modified SHUTi (SHUTi modified for Black women) (Active Comparator): The CBT-I instrument tailored for Black women.
  Interventions: Behavioral: modified SHUTi (i.e., SHUTi-BWHS)

INTERVENTIONS:
Behavioral: SHUTi — A woman assigned to SHUTi receives access to an online program that includes 6 interactive sessions that are designed to be reviewed over a period of about 8 weeks. The online sessions include videos and written material that give information about factors that affect sleep, changes that might help sleep patterns, and how to make those changes. Each session takes about 45 to 60 minutes to complete. During and between sessions, the participant fills out sleep diaries to gather information about daily sleep patterns. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health as well as sleep diaries. Time 1 is just before starting the first session of the SHUTi program. Time 2 is about 9 weeks later and Time 3 is about six months after that. The questionnaires will be used to assess the effect of the online program on the participant's sleep and health.
  Other Names: web-based cognitive-behavioral therapy for insomnia (CBT-I)
  Arms: SHUTi (Sleep Healthy Using the Internet)
Behavioral: modified SHUTi (i.e., SHUTi-BWHS) — A woman assigned to modified SHUTi (i.e., to SHUTi-BWHS) receives access to an online program that includes 6 interactive sessions that are designed to be reviewed over a period of about 8 weeks. The online sessions include videos and written material that give information about factors that affect sleep, changes that might help sleep patterns, and how to make those changes. Each session takes about 45 to 60 minutes to complete. During and between sessions, the participant fills out sleep diaries to gather information about daily sleep patterns. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health as well as sleep diaries. Time 1 is just before starting the first session of the modified SHUTi program. Time 2 is about 9 weeks later and Time 3 is about six months after that. The questionnaires will be used to assess the effect of the online program on the participant's sleep and health.
  Other Names: web-based CBT-I tailored for Black women
  Arms: modified SHUTi (SHUTi modified for Black women)
Behavioral: Patient education — A woman assigned to patient education receives access to a website that provides detailed information on habits and environments that may help or hinder sleep. The site can be visited as often as desired. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health, as well as sleep diaries to gather information about her daily sleep pattern. Time 1 is just before first logging into the sleep information website. Time 2 is about 9 weeks later and Time 3 is six months after that. The questionnaires will be used to assess the effect of the sleep information program on the participant's sleep and health.
  Other Names: sleep hygiene
  Arms: Patient education (sleep hygiene)

SUMMARY:
Black women are at a higher risk of developing insomnia than other women and insomnia has profound adverse physical and psychological health consequences. There is an internet-delivered treatment program for insomnia that has been shown to be effective in White individuals but there is little evidence of the effectiveness of this treatment among Black women. The goal of this study is to conduct a comparative effectiveness trial of three online insomnia therapies after a 6 month follow-up period--a cognitive behavioral therapy for insomnia (CBT-I) called SHUTi (Sleep Healthy Using the Internet), SHUTi modified for Black women (SHUTi-BWHS), and patient education (PE) (usual treatment). This study aims to provide the much needed evidence to help Black women make informed decisions regarding treatment for their insomnia.

DETAILED DESCRIPTION:
Eligible Black Women's Health Study (BWHS) participants who completed the Insomnia Severity Index(ISI) on the 2015 BWHS questionnaire with a score compatible with insomnia disorder will be randomly selected to receive information that will inform them of the opportunity to participate in a free program designed to address their sleep problems. They will then be directed to an Insomnia Study Website which will provide information about the study and directions on how to complete an online screening questionnaire for those interested in participating. Reminders will be sent to these selected women to encourage participation.

Once interested women submit the screening questionnaire, an internal assessment will be carried out to see if potential participants are eligible. Those determined to be ineligible will be sent a thank you letter and informed that they were not selected for this trial. Those who meet the qualifications for the study will be directed to the informed consent form with a note indicating that a member of the study team will call them within several days at a time they indicated would be convenient for them. The study team member will then call each eligible subject and review with her, over the phone, each section of the consent form. A verbal acknowledgement of consent, or non-consent, will be recorded in the study database.

Once women have been verbally consented, they will be instructed on the use of the web programs and, completion of online sleep logs. Privacy concerns will be addressed. Pre-intervention, post-intervention, and 6-month assessment questionnaires, including the Insomnia Severity Index (ISI) will be administered pre-intervention (Time 1), post-intervention 9 weeks after Time 1 (Time 2), and 6 months later (Time 3). After the pre-intervention questionnaires and sleep logs are completed, participants will be informed of their treatment which was selected at random from the three online treatments: SHUTi -BWHS, SHUTi, and patient education (PE) (also called sleep hygiene or sleep information). The PE group will use a website that discusses ways to improve behaviors and environments that can affect sleep. This material is also included in the other 2 treatments but is presented in a different way. Participants using the PE website may log in as often as they like for as long as they like. Participants randomized to SHUTi-BWHS or SHUTi will use a web program that has six modules called Cores. Participants will log in to the six modules of their assigned treatment program over an 8-week period. Cores are completed one at a time in order. Each Core is expected to take 45 to 60 minutes to complete. Each Core contains information and exercises designed to help change behaviors and thoughts that can contribute to sleep problems.

Nine weeks after completing the initial pre-intervention questionnaire, all participants will be asked to complete another questionnaire about their sleep and health, which includes the ISI, and also to complete 10 sleep diaries. Six months later, participants will be asked again to complete a questionnaire that includes the ISI, followed by completion of 10 sleep diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Participants in the Black Women's Health Study (BWHS) with clinically elevated symptoms of insomnia previously reported on a BWHS questionnaire.
2. Access to a computer or tablet and internet access

Exclusion Criteria:

1. Intention to change use pattern of prescribed or over-the-counter sleep aid
2. 1 or more untreated sleep disorders
3. Employed in a position where sleep restriction may endanger others
4. Active shift work employment
5. Untreated, current, and/or severe psychiatric condition
6. Consume 14 or more alcoholic drinks/week
7. Unstable or acute medical condition

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants in the Black Women's Health Study who have reported symptoms of insomnia on the 2015 BWHS follow-up questionnaire
Enrollment: 333 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Rosenberg, ScD, Principal Investigator — Senior Epidemiologist, Professor of Epidemiology; Eric S Zhou, PhD, Principal Investigator — Division of Sleep Medicine, Harvard Medical School
Locations (1):
- Slone Epidemiology Center at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou ES, Ritterband LM, Bethea TN, Robles YP, Heeren TC, Rosenberg L. Effect of Culturally Tailored, Internet-Delivered Cognitive Behavioral Therapy for Insomnia in Black Women: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jun 1;79(6):538-549. doi: 10.1001/jamapsychiatry.2022.0653. PMID 35442432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1010 completed the eligibility questionnaire. 490 were excluded for not meeting criteria and 187 declined to participate. The remaining 333 were randomized into one of the three trial arms.
Groups:
- Patient Education (Sleep Hygiene, Usual Care): A web-based program that presents ways to improve behaviors and environments that can affect sleep.
  Patient education: A woman assigned to patient education receive access to a website that provides detailed information on habits and environments that may help or hinder sleep. The site can be visited as often as desired. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health, as well as sleep diaries to gather information about her daily sleep pattern. Time 1 is just before first logging into the sleep information website. Time 2 is about 9 weeks later and Time 3 is six months after that. The questionnaires will be used to assess the effect of the sleep information program on the participant's sleep and health.
- SHUTi (Sleep Healthy Using the Internet): SHUTi (Sleep Healthy Using the Internet) is web-based cognitive-behavioral therapy instrument for insomnia (CBT-I)
  SHUTi: A woman assigned to SHUTi receives access to an online program that includes 6 interactive sessions that are designed to be reviewed over a period of about weeks. The online sessions include videos and written material that give information about factors that affect sleep, changes that might help sleep patterns, and how to make those changes. Each session takes about 45 to 60 minutes to complete. During and between sessions, the participant fills out sleep diaries to gather information about daily sleep patterns. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health as well as sleep diaries. Time 1 is just before starting the first session of the SHUTi program. Time 2 is about 9 weeks later and Time 3 is about six months after that. The questionnaires will be used to assess the effect of the online program on the participant's sleep and health.
Period: Baseline
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Started | 115 | 108 | 110
Completed | 113 | 85 | 100
Not Completed | 2 | 23 | 10
Period: Post -Intervention (9 Weeks)
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Started | 113 | 85 | 100
Completed | 112 | 79 | 93
Not Completed | 1 | 6 | 7
Period: Long-term Follow-up (6 Months)
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Started | 112 | 79 | 93
Completed | 112 | 79 | 93
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Modified SHUTi (SHUTi Modified for Black Women): The CBT-I instrument tailored for Black women.
  Modified SHUTi (i.e., SHUTi-BWHS): A woman assigned to modified SHUTi (i.e., to SHUTi-BWHS) receives access to an online program that includes 6 interactive sessions that are designed to be reviewed over a period of 6 to 8 weeks. The online sessions include videos and written material that give information about factors that affect sleep, changes that might help sleep patterns, and how to make those changes. Each session takes about 45 to 60 minutes to complete. During and between sessions, the participant fills out sleep diaries to gather information about daily sleep patterns. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health as well as sleep diaries. Time 1 is just before starting the first session of the modified SHUTi program. Time 2 is about 9 weeks later and Time 3 is about six months after that. The questionnaires will be used to assess the effect of the online program on the participant's sleep and health.
- Total: Total of all reporting groups
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women) | Total
Number analyzed (Participants) | 115 | 108 | 110 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (7.7) | 59.9 (8.0) | 59.6 (8.4) | 59.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 108 | 110 | 333
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 115 | 108 | 110 | 333
Region of Enrollment [Number; unit: participants]
  United States | 115 | 108 | 110 | 333
Weekly alcohol consumption [Mean (Standard Deviation); unit: drinks per week] | 1.2 (2.1) | 1.8 (2.6) | 1.1 (1.9) | 1.4 (2.2)
Smoking history [Number; unit: percent of participants]
  Current | 4 | 9 | 5 | 6
  Past | 24 | 17 | 29 | 23
  Never | 71 | 74 | 66 | 71
Body Mass Index (BMI= kg/m^2) [Number; unit: percent of participants]
  <25 | 16 | 23 | 30 | 23
  25-29 | 27 | 26 | 23 | 25
  30 or greater | 51 | 47 | 40 | 46
  Unknown | 6 | 4 | 7 | 6
Insomnia Severity Index [Mean (Standard Deviation); unit: score on a scale] — The Insomnia Severity Index (ISI) is a measure of symptoms of insomnia. The range of scores is 0 to 28. A score less than 8 indicates no clinically significant symptoms of insomnia. A score of 8 - 14 indicates some .symptoms of insomnia. A score of 15 - 28 indicates clinical insomnia. Higher scores indicate worse insomnia.
  score on a scale | 19.2 (0.3) | 18.3 (0.4) | 18.7 (0.4) | 18.8 (0.2)
Sleep Onset Latency [Mean (Standard Deviation); unit: minutes] | 41.6 (2.6) | 47.5 (2.7) | 38.0 (2.7) | 42.3 (1.6)
Total Sleep Time [Mean (Standard Deviation); unit: hours] | 5.7 (0.1) | 5.7 (0.1) | 6.0 (0.1) | 5.8 (0.1)
Sleep Efficiency [Mean (Standard Deviation); unit: percent] — Sleep Efficiency (SE) is the percent of time bed asleep. Sleep efficiency of at least 85% is desirable.
  percent | 72.7 (1.1) | 70.9 (1.1) | 73.1 (1.1) | 72.2 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Difficulties Assessed by the Insomnia Severity Index
Description: A change in sleep difficulties will be assessed by the change in the ISI (Insomnia Severity Index) score. The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the past month. The specific items evaluate the severity of difficulties with sleep onset, sleep maintenance, and early morning awakening; sleep dissatisfaction; interference of sleep problems with daytime functioning; noticeability of sleep difficulties by others; and distress caused by sleep difficulties. A 5-point Likert scale (0 = none; 4 = very severe) is used to rate each item, with total scores ranging from 0 to 28. A higher total score indicates more severe sleep difficulties.
Time Frame: Time 1 (baseline), Time 3 (6 months after expected completion of program)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Patient Education (Sleep Hygiene, Usual Care): A web-based program that presents ways to improve behaviors and environments that can affect sleep.
  Patient Education: A woman assigned to Patient Education receives access to a website that provides detailed information on habits and environments that may help or hinder sleep. The site can be visited as often as desired. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health, as well as sleep diaries to gather information about her daily sleep pattern. Time 1 is just before first logging into the sleep information website. Time 2 is about 9 weeks later and Time 3 is six months after that. The questionnaires will be used to assess the effect of the sleep information program on the participant's sleep and health.
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Number analyzed (Participants) | 112 | 79 | 93
score on a scale | -3.6 (0.5) | -10.0 (0.6) | -9.3 (0.6)

2. Secondary Outcome: Change in Sleep Onset Latency (SOL)
Description: SOL is the amount of time it takes to fall asleep measured in minutes.
Time Frame: Time 1 (baseline), Time 3 (6 months after expected completion of program)
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Number analyzed (Participants) | 112 | 79 | 93
Minutes | -7.0 (2.7) | -20.2 (3.0) | -17.7 (2.8)

3. Secondary Outcome: Change in Wake After Sleep Onset (WASO)
Description: WASO measures time awake after falling asleep measured in minutes.
Time Frame: Time 1 (baseline), Time 3 (6 months after expected completion of program)
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Number analyzed (Participants) | 112 | 79 | 93
minutes | -7.2 (2.9) | -17.6 (3.3) | -19.7 (3.1)

4. Secondary Outcome: Change in Total Sleep Time (TST)
Description: TST is the amount of time spent asleep in bed, measured in minutes and then converted to hours. Total sleep time is calculated by subtracting SOL (Sleep Onset Latency, WASO (Wake After Sleep Onset) and EMA (Early Morning Arise) from total time in bed (TIB).
Time Frame: Time 1 (baseline), Time 3 (6 months after expected completion of program)
Measure: Mean (Standard Error); unit: hours
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Number analyzed (Participants) | 112 | 79 | 93
hours | 0.5 (0.1) | 0.8 (0.1) | 0.3 (0.1)

5. Secondary Outcome: Change in Sleep Efficiency (SE)
Description: Change in Sleep Efficiency (SE). SE is the change in the percentage of time spent asleep while in bed. SE is calculated by dividing the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes) times 100.
Time Frame: Time 1 (baseline), Time 3 (6 months after expected completion of program)
Measure: Mean (Standard Error); unit: percent
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Number analyzed (Participants) | 112 | 79 | 93
percent | 4.3 (1.1) | 12.3 (1.2) | 11.4 (1.1)

6. Secondary Outcome: Completion of All 6 Cores/Modules
Description: The percentage of participants in the SHUTi and modified SHUTI arms who completed all six cores/modules during the study
Time Frame: Time 3 (6 months after expected completion of program)
Population: Only participants in the SHUti and the modified SHUTi arms used the cores/modules, so this outcome was not measured in the usual care arm.
Measure: Number; unit: percentage of participants
Arm/Group | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
Number analyzed (Participants) | 70 | 86
percentage of participants | 64.8 | 78.2

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Modified SHUTi (SHUTi Modified for Black Women): The CBT-I instrument tailored for Black women.
  Modified SHUTi (i.e., SHUTi-BWHS): A woman assigned to modified SHUTi (i.e., to SHUTi-BWHS) receives access to an online program that includes 6 interactive sessions that are designed to be reviewed over a period of of about 8 weeks. The online sessions include videos and written material that give information about factors that affect sleep, changes that might help sleep patterns, and how to make those changes. Each session takes about 45 to 60 minutes to complete. During and between sessions, the participant fills out sleep diaries to gather information about daily sleep patterns. At 3 different times, the woman is asked to fill out questionnaires about her sleep and health as well as sleep diaries. Time 1 is just before starting the first session of the modified SHUTi program. Time 2 is about 9 weeks later and Time 3 is about six months after that. The questionnaires will be used to assess the effect of the online program on the participant's sleep and health.
Arm/Group | Patient Education (Sleep Hygiene, Usual Care) | SHUTi (Sleep Healthy Using the Internet) | Modified SHUTi (SHUTi Modified for Black Women)
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/108 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/108 | 0/110
Other Adverse Events (participants affected / at risk) | 0/115 | 0/108 | 0/110

LIMITATIONS AND CAVEATS:
The study sample, comprised entirely of Black women who have not previously been studied, are of a higher socioeconomic background than US Black women as a whole. However, participants lived in a wide range of settings across the country, encountering a variety of circumstances that might impair sleep.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03613519/Prot_SAP_000.pdf